CLINICAL TRIAL: NCT03220555
Title: Efficacy of a Cold, Vibration, and Distraction Based Medical Device on the Prevention of Health Care Induced Pediatric Pain: a Comparative, Controlled, Randomized and Multicentric Study
Brief Title: Efficacy of the Buzzy® Device on the Prevention of Health Care Induced Pediatric Pain in a Vaccination Center
Acronym: DOLVAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC17_0035
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Intravenous Injections; Vaccination
Keywords: Buzzy; anesthetic cream; pediatric; pain; venipuncture; vaccination; vibration; cold; distraction; vaccination center
MeSH Terms: conditions — Pain; Common Cold | interventions — Lidocaine; Prilocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buzzy® device (Experimental): Just before the vaccination or venipuncture the device will be applied on the selected site during 30 seconds and then it will be moved 5 cm above the selected site to make the injection or the puncture. The child will choose if he wants to use the cooling system.
  Interventions: Device: Buzzy® device
- EMLAPATCH (lidocaine, prilocaine) (Active Comparator): The patch will be applied during 1 hour to 1 hour and half before the vaccination or venipuncture, on the selected site. After 1 hour to 1 hour and half, it will be removed and the injection or the puncture will be made on the selected site.
  Interventions: Drug: EMLAPATCH (lidocaine, prilocaine)

INTERVENTIONS:
Device: Buzzy® device — Just before the vaccination or venipuncture the device will be applied on the selected site during 30 seconds and then it will be moved 5 cm above the selected site to make the injection or the puncture. The child will choose if he wants to use the cooling system.
  Arms: Buzzy® device
Drug: EMLAPATCH (lidocaine, prilocaine) — The patch will be applied during 1 hour to 1 hour and half before the vaccination or venipuncture, on the selected site. After 1 hour to 1 hour and half, it will be removed and the injection or the puncture will be made on the selected site.
  Arms: EMLAPATCH (lidocaine, prilocaine)

SUMMARY:
In vaccination centers, venipunctures and vaccinations are sources of pain and anxiety in pediatric patients. Prior painful experiences can reduce the acceptance of later health care, hence making it more difficult for both patients and nurses.

The topical anesthetic cream (lidocaine, prilocaine) and the non-pharmacological (distraction and relaxation) interventions which are usually used for prevention of procedural pain impose certain constraints on families and on vaccination centers.

A distraction and local anesthesia (cold and vibration) based medical device (Buzzy®) could overcome these constraints and could be an interesting alternative for healthcare management in vaccination centers and, in a broader perspective, in other medical services.

Research on this device has been scarce to date. Three of them have shown an efficacy of Buzzy® in comparison to the absence of prevention of vaccination and venipuncture induced pain. An ongoing study will assess the Buzzy® device in comparison to a topical anesthetic cream, but will be set in an emergency department context. To date, no study has compared Buzzy® to topical anesthetic cream on healthy children in a vaccination center.

The research team has formulated the following hypothesis: the Buzzy® device will allow to get a not lower or an equivalent level of pain compared to the level of pain obtained with the usual topical anesthetic cream. The aim of this study is to evaluate the efficacy of the device Buzzy® on vaccination and venipuncture induced pain in a vaccination center.

ELIGIBILITY:
Inclusion Criteria:

Any child who:

* requires a venipuncture or a vaccination in a vaccination center
* is 4 to 15 years old
* is affiliated to the public social security
* speaks French or is assisted by an translator in the language of the child
* has given his oral consent and whose parents have given it

Exclusion Criteria:

Any child who:

* suffers from sickle cell anemia
* has a contraindication to use lidocaine patch
* requires a Bacille de Calmette et Guérin (BCG) vaccine or tuberculin test
* takes part in another research
* has already participated to this study for another nursing care.
* refused to participate or whose parents refused
* has neurological or psychiatric disorders
* has a nerve damage or an abrasion of the skin in terms of puncture or injection area.
* under trusteeship or guardianship (unaccompanied foreign minors).

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Faces Pain Scale revised (FPS-r) for children | Day 0
  Pain will be assessed by child using the FPS-r. FPS-r is a tool which has been validated and has been shown to be reliable in intercultural children and adolescents population (4 to 17 years).

SECONDARY OUTCOMES:
Faces Pain Scale revised (FPS-r) for parents | Day 0
  Pain will be assessed by a parent using the FPS-r. FPS-r is a tool which has been validated and has been shown to be reliable in intercultural children and adolescents population (4 to 17 years).
Differential cost of the two strategies compared to the differential pain | Day 0
  Differential cost of the two strategies compared to the differential pain, self-reported by children with the FPS-r. Cost assessment of the two strategies will be made by a micro-costing analysis. The parameters analyzed will be : the strategy used (Buzzy® device or EMLAPATCH), the nurses' time and the time spent by child in the vaccination center. This parameters will be aggregated and will be presented in the form of a cost-effectiveness differential ratio and acceptability curves.

CONTACTS AND LOCATIONS:
Overall Officials: Lescop Katia, IDE, Principal Investigator — Nantes University Hospital
Locations (3):
- France (3):
  - La Roche sur Yon University Hospital, La Roche-sur-Yon
  - Le Mans University Hospital, Le Mans
  - Nantes University Hospital, Nantes